CLINICAL TRIAL: NCT04353778
Title: Effects of Vagal Dysfunction on Gastrointestinal and Inflammatory Pathways in HIV
Acronym: EVA
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jessica Robinson-Papp, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 18-2812; 1R01DK122853-01A1 (NIH)
Record Dates: First submitted 2020-04-17; First posted 2020-04-20 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: HIV; Non-HIV; Vagus Nerve Dysfunction
Keywords: Small intestinal bacterial overgrowth; People living with HIV; HIV-associated autonomic neuropathy; Distal symmetric polyneuropathy
MeSH Terms: interventions — Pyridostigmine Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- PLWH (No Intervention): People living with HIV (HIV)
- Healthy Controls (No Intervention): Healthy controls who do not have HIV
- Pyridostigmine (Active Comparator): PLWH on pyridostigmine 30mg PO TID
  Interventions: Drug: Pyridostigmine
- Placebo (Placebo Comparator): PLWH on placebo
  Interventions: Drug: Placebos
- nVNS (Other): PLWH to undergo non-invasive vagal nerve stimulation
  Interventions: Procedure: non-invasive vagal nerve stimulation

INTERVENTIONS:
Drug: Pyridostigmine — Eight weeks of low-dose pyridostigmine
  Arms: Pyridostigmine
Drug: Placebos — matching placebo x 8 weeks
  Arms: Placebo
Procedure: non-invasive vagal nerve stimulation — stimulation of the vagus nerve
  Other Names: nVNS
  Arms: nVNS

SUMMARY:
The study team's prior research has shown that dysfunction of a specific nerve, called the vagus nerve, is associated with small intestinal bacterial overgrowth (SIBO), and that SIBO is associated with signs of inflammation in the blood of people living with HIV (PLWH). This research will explore pathways linking vagal dysfunction to inflammation in HIV, focusing on the gastrointestinal tract, and study whether a medication called pyridostigmine and stimulation of the vagus nerve are beneficial therapies.

DETAILED DESCRIPTION:
Objectives Aim 1: To elucidate mechanisms linking VD, SIBO and chronic inflammation in PLWH. PLWH (N=150) will undergo autonomic function tests (AFTs) for VD, hydrogen/methane breath testing (HBT) for SIBO, Wireless Motility Capsule (WMC, SmartPill) testing for GI transit times and pH measurements, blood draw for quantification of inflammatory mediators, and collection of stool samples and oral swabs for characterization of the GI microbiome.

Hypothesis 1a (primary): The relationship between VD and SIBO in HIV is mediated by prolonged small bowel transit time (SBTT) and hypochlorhydria.

Hypothesis 1b (exploratory): There is an additional pathway linking VD and elevated IL-6 in PLWH which is independent of SIBO and bacterial translocation.

Aim 2: To determine whether the relationship between VD and SIBO is modified by the presence of HIV-infection. HIV-infection results in disruption of the GI mucosal barrier,5 which could make PLWH more vulnerable to adverse GI effects of VD. HIV-uninfected controls (N=100), age and gender matched to the PLWH from Aim 1, will undergo the same assessment as the PLWH. The study team will test for effect modification of the VD-SIBO relationship by HIV status, using logistic regression to examine the interaction between VD and HIV.

Aim 3: To establish vagal pathways as a viable treatment target for individuals with well-controlled HIV. PLWH with VD, SIBO and/or prolonged SBTT (N=96) will be identified from the Aim 1 cohort. The first 86 eligible patients will be randomized to 8 weeks of pyridostigmine versus placebo; the remaining 10 will receive 8 weeks of open-label noninvasive vagal nerve stimulation (nVNS) to assess feasibility. All patients will then be retested (AFTs, HBT, SmartPill, blood draw, stool samples and oral swabs).

Hypothesis 3a (primary): Eight weeks of low-dose pyridostigmine (30mg PO TID) will reduce SIBO as compared to placebo in PLWH. Hypothesis 3b (exploratory): Non-invasive VNS is safe, well tolerated and acceptable to PLWH.

ELIGIBILITY:
Inclusion Criteria :

* Greater than or equal to18 years old (18 to 64 Years, 65 Years and Over)
* Documentation of HIV-1 infection
* Stable CART for greater or equal to 3 months
* HIV-1 viral load <100 copies/ml (within 3m)
* No diagnosis known to cause autonomic or GI dysfunction other than HIV (e.g. Parkinson's disease, diabetes, peptic ulcer disease, infectious diarrhea)
* Willing to refrain from nicotine use for 24h prior to all testing
* No contraindication to autonomic testing (e.g. uncontrolled glaucoma, heart rate not under sinus control)
* No medications with significant autonomic or GI effects (e.g. sympathomimetics, prokinetics, anti-diarrheals, antibiotics)
* Urine test negative for stimulants and opiates/opioids and pregnancy test (if applicable)

Exclusion Criteria:

* Dysphagia to food or pills
* Known or suspected obstructive disease of the GI tract (e.g. bezoar, strictures, fistulae, physiologic GI obstruction)
* GI surgery within 3m, Crohn's disease, diverticulitis, any electromechanical medical device (e.g. pacemaker, infusion pump).
* Contraindication to pyridostigmine (e.g. mechanical intestinal or urinary obstruction, hypersensitivity to pyridostigmine, cardiac arrhythmias, asthma, chronic obstructive pulmonary disease); use of pyridostigmine within the past 6m.
* History of intracranial aneurysm/hemorrhage, brain tumor, abnormal neck anatomy, or implants or metal hardware near site of stimulation; exposure to VNS within the past 6m.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Small bowel transit time (SBTT) | 8 weeks
  Small bowel transit time (SBTT) measured by wireless motility capsule (wmc, smartpill)
Gastric pH measurement | 8 weeks
  Gastric pH measurement measured by wireless motility capsule (wmc, smartpill)
Hydrogen/methane breath testing (hbt) | 8 weeks
  hydrogen/methane breath testing (hbt) to measure small intestinal bacterial overgrowth
IL6 measurement [Time Frame: 5 years] | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Robinson-Papp, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: CSR
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Anyone who wishes to access the data. Data will be published.

REFERENCES:
- [Background] Robinson-Papp J, Nmashie A, Pedowitz E, George MC, Sharma S, Murray J, Benn EKT, Lawrence SA, Machac J, Heiba S, Kim-Schulze S, Navis A, Roland BC, Morgello S. The effect of pyridostigmine on small intestinal bacterial overgrowth (SIBO) and plasma inflammatory biomarkers in HIV-associated autonomic neuropathies. J Neurovirol. 2019 Aug;25(4):551-559. doi: 10.1007/s13365-019-00756-9. Epub 2019 May 16. PMID 31098925
- [Background] Carod-Artal FJ. Infectious diseases causing autonomic dysfunction. Clin Auton Res. 2018 Feb;28(1):67-81. doi: 10.1007/s10286-017-0452-4. Epub 2017 Jul 20. PMID 28730326
- [Background] Robinson-Papp J, Nmashie A, Pedowitz E, Benn EKT, George MC, Sharma S, Murray J, Machac J, Heiba S, Mehandru S, Kim-Schulze S, Navis A, Elicer I, Morgello S. Vagal dysfunction and small intestinal bacterial overgrowth: novel pathways to chronic inflammation in HIV. AIDS. 2018 Jun 1;32(9):1147-1156. doi: 10.1097/QAD.0000000000001802. PMID 29596112
- [Background] Paulon E, Nastou D, Jaboli F, Marin J, Liebler E, Epstein O. Proof of concept: short-term non-invasive cervical vagus nerve stimulation in patients with drug-refractory gastroparesis. Frontline Gastroenterol. 2017 Oct;8(4):325-330. doi: 10.1136/flgastro-2017-100809. Epub 2017 May 24. PMID 29067158
- [Background] Lerman I, Hauger R, Sorkin L, Proudfoot J, Davis B, Huang A, Lam K, Simon B, Baker DG. Noninvasive Transcutaneous Vagus Nerve Stimulation Decreases Whole Blood Culture-Derived Cytokines and Chemokines: A Randomized, Blinded, Healthy Control Pilot Trial. Neuromodulation. 2016 Apr;19(3):283-90. doi: 10.1111/ner.12398. Epub 2016 Mar 15. PMID 26990318
- [Background] Tarn J, Legg S, Mitchell S, Simon B, Ng WF. The Effects of Noninvasive Vagus Nerve Stimulation on Fatigue and Immune Responses in Patients With Primary Sjogren's Syndrome. Neuromodulation. 2019 Jul;22(5):580-585. doi: 10.1111/ner.12879. Epub 2018 Oct 17. PMID 30328647